CLINICAL TRIAL: NCT06050200
Title: Comparison of Three Methods of Inducing Liver Hypertrophy Before Resection - a Randomized Controlled Trial
Brief Title: TANGO-LIVER Three Arm Nuclear Growth Observation in Liver Surgery
Acronym: TANGO-LIVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABM24
Record Dates: First submitted 2023-08-31; First posted 2023-09-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Liver Metastases; Liver Cancer; Liver Neoplasms; Liver Metastasis Colon Cancer
Keywords: liver metastases; liver cancer; liver neoplasms; portal vein embolisation; liver venous deprivation; PVE; LVD; Associating Liver Partition and Portal vein Ligation for Staged hepatectomy; ALPPS; liver resection; mebrofenin scintigraphy; liver surgery
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional randomized study. Patients will be randomly assigned to three groups in a 12:71:71 ratio: PVE, LVD and ALPPS groups, respectively.
  Randomization will be performed directly after recruitment.
Who Masked: Participant, Investigator
Masking Description: The Investigator performing statistical analysis will blinded to which study group the patient was assigned to.
  The patient will not be aware which of the two radiological methods (PVE or LVD) was performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PVE (Active Comparator): Portal Vein Embolisation Patients in this group will undergo embolisation of branch of portal vein (interventional radiological procedure)
  Interventions: Procedure: PVE
- LVD (Active Comparator): Liver Venous Deprivation Patients in this group will undergo simultaneous embolization of branch of the portal vein and one or two hepatic veins (interventional radiological procedure)
  Interventions: Procedure: LVD
- ALPPS (Experimental): Associating Liver Partition and Portal vein Ligation for Staged hepatectomy: Patients in this group will undergo surgical ligation of portal vein branch with partial liver transection (surgical procedure)
  Interventions: Procedure: ALPPS

INTERVENTIONS:
Procedure: PVE — The procedure is performed under general anesthesia. Ultrasound-guided percutaneous, transhepatic puncture of the branch of the portal vein is performed and a vascular sheath is inserted on the guidewire. A system of catheters and guidewires is inserted through the sheath. Embolization is performed using a homogeneous mixture of Glubran 2 glue and Lipiodol (volume ratio 1:8-1:9). After filling the entire volume of the branch of the portal vein, all catheters, guidewires and the vascular sheaths are removed. A dressing is left over the access site and removed the next day. After treatment the patient is given analgesics and antipyretics if necessary.
  Other Names: portal vein embolization
  Arms: PVE
Procedure: LVD — The procedure is performed under general anesthesia. Ultrasound-guided percutaneous, transhepatic puncture of the branch of the portal vein is performed and a vascular sheath is inserted on the guidewire. A system of catheters and guidewires is inserted through the sheath. A similar puncture of the hepatic vein or veins is then performed; sometimes with access via the internal jugular vein. Embolization of the portal branch is performed using a homogeneous mixture of Glubran 2 glue and Lipiodol (volume ratio 1:8-1:9). Embolization of the right hepatic vein or veins begins with the insertion of a vascular plug (Amplatzer) approx. 2 cm from the confluence of the vein(s). The remaining part of the hepatic vein(s) is then filled with a homogeneous mixture of histacryl glue and Lipiodol (volume ratio 1:1).
  A dressing is left over the access site and removed the next day; patient is given analgesics and antipyretics if necessary.
  Other Names: liver venous deprivation
  Arms: LVD
Procedure: ALPPS — The ALPPS procedure will be performed in the operating theatre, under general anesthesia, preferably using a minimally invasive (laparoscopic) technique.
  The procedure consists of surgical ligation or clipping of the branch of the portal vein with a vascular clip and in partial transection of the parenchyma at the plane of the future resection planned in the second stage (partial transection, approx. 75% of the transection plane).
  Other Names: Associating Liver Partition and Portal vein Ligation for Staged hepatectomy
  Arms: ALPPS

SUMMARY:
Liver resection is the treatment of choice in patients with malignant liver lesions. Unfortunately, the surgery is not always an option, as in same patients the future remnant liver (FRL) is too small to supply all the functions. Therefore, some additional methods have been proposed to increase the size of the FRL.

The aim of this study is to compare the efficacy and safety of three methods of increasing the future remnant liver - Portal Vein Embolization (PVE) - embolization of one of the portal branches; Liver Vein Deprivation (LVD) - embolization both of the portal branch as well as the hepatic vein; and partial ALPPS (Associating Liver Partition and Portal vein Ligation for Staged hepatectomy) - ligation of portal vein branch with partial liver transection.

The efficacy of those three methods will be assessed both by analyzing the volumetric increase (by computer tomography scans) and by functional increase (by 99mTc-mebrofenin scintigraphy). Functional assessment of the liver hypertrophy seems to be of crucial importance, as some of the previous studies suggest that there might be a significant discrepancy in the increase of size comparing to the increase of function.

This is a prospective, interventional randomized study. The study group (154 patients) will consist of patients being considered as candidates for major hepatic resection, after inducing hypertrophy of the future remnant liver.

The primary study hypothesis is greater efficacy of ALPPS in preparing patients for large hepatic resection by inducing hypertrophy of the future remnant liver, as compared both to PVE and LVD.

In case of unsuccessful induction of hypertrophy by the embolization techniques, patients may be qualified to rescue ALPPS procedure.

Primary end-point:

Percentage of patients with successful resection (patients, who gained sufficient increase of the FRL to proceed to the liver resection) with no post-surgical 90-day mortality.

Secondary end-points:

1. the rate and degree of volume increase in different groups
2. the rate and degree of functional increase in different groups
3. CCI index and complication rate >=3 degree according to the Clavien-Dindo classification after the first stage of treatment
4. CCI index and complication rate >=3 degree according to the Clavien-Dindo classification after the second stage of treatment
5. overall duration of hospital stay

Patient will be randomly assigned to the three study groups. All patients will undergo an abdominal contrast enhanced computed tomography and 99mTc-mebrofenin scintigraphy prior to the first stage of treatment. During the first stage of treatment, patients will undergo, according to their group:

1. Embolization of portal vein branch (PVE, portal vein embolization)
2. Embolization of both portal vein branch and hepatic vein (LVD, liver venous deprivation)
3. Partial ALPPS (Associating Liver Partition and Portal vein Ligation for Staged hepatectomy) - ligation of portal vein branch with partial liver transection, preferentially by laparoscopic technique Computed tomography scans and scintigraphy will be repeated at day 7, 14 and 21 after the first stage of treatment. The second stage of treatment, the liver resection, will be performed after achievement of sufficient mebrofenin clearance rate (>=2,69%/min/m2). In case of failure to reach the desired clearance rate, the measurements will be continued every 7 days up to day 42. In case of uncertainty and discrepancy between the volumetric assessment in the computed tomography scan and the mebrofenin scintigraphy, it will be allowed to proceed to stage two (partial hepatectomy) after joint consultation of at least 3 hepatobiliary surgeons, 1 radiologist and 1 nuclear medicine specialist. Routine blood tests will be performed according to the standard procedure in the Department, depending on the patient clinical status. An additional blood sample will be collected from patients (after receiving and additional informed consent from the patient) and will be stored in the biobank.

All patients will be monitored for surgical and 90-day complications. The volume increase after first stage of treatment, the functional increase after first stage of treatment, percentage of patients successfully proceeding to the second stage of treatment and complication rate will be calculated.

The percentage of patients with complications >= 3 degree in Clavien-Dindo classification and CCI index for each patient will be calculated.

Furthermore, the blood test results will be assessed to search for associations with patients' outcomes. Any possible differences in terms of baseline patients characteristics between groups will be addressed.

Statistical analysis will be performed using U Mann-Whitney test, exact Fisher's test, logistic regression, general linear models, Kaplan-Meier method and log-rank test. All three groups will be assessed in terms of occurrence of primary and secondary end-points.

DETAILED DESCRIPTION:
Liver resection is the treatment of choice in patients with malignant liver lesions. Unfortunately, the surgery is not always an option, as in same patients the future remnant liver (FRL) is too small to supply all the functions. Therefore, some additional methods have been proposed to increase the size of the FRL. Among the most widely used ones are: Portal Vein Embolization (PVE) - embolization of one of the portal branches; Liver Vein Deprivation (LVD) - embolization both of the portal branch as well as the hepatic vein and partial ALPPS (Associating Liver Partition and Portal vein Ligation for Staged hepatectomy) - ligation of portal vein branch with partial liver transection.

However, for the time being none of this methods has been proven to provide superior results in comparison to other, and all of them are widely used in different centers. Most of the previously published papers were retrospective in nature and as for now there was no randomized trial conducted to compare all three of them. What is more, most of the previously published papers focused on the volumetric increase, based solely on the computed tomography analysis. The most important is however the functional increase, not the increase in size. The functional increase can be assessed in the 99mTc-mebrofenin scintigraphy, which enables to assess the liver function in a chosen part of the liver.

Some of the previously published papers indicate that there might be a significant discrepancy in the increase of size comparing to the increase of function, which is critically important in the clinical practice.

The aim of this study is to compare the efficacy and safety of three methods of increasing the future remnant liver - PVE, LVD and ALPPS in patients in whom liver resection is considered.

METHODS:

This is a prospective, interventional randomized study. Patients will be randomly assigned to three groups in a 12:71:71 ratio: PVE, LVD and ALPPS groups, respectively.

Randomization will be performed directly after recruitment. The study group will consist of patients being considered as candidates for major hepatic resection, after inducing hypertrophy of the future remnant liver.

Inclusion criteria:

1. age >= 18 years
2. patients qualified for liver resection
3. future remnant liver <30% of standard liver volume
4. written informed consent

Exclusion criteria:

1. liver cirrhosis
2. pregnancy
3. poor general health status or comorbidities excluding general anesthesia or hepatic resection
4. contraindications to iodine contrast agents

Hypothesis and study group:

The primary study hypothesis is greater efficacy of ALPPS in preparing patients for large hepatic resection by inducing hypertrophy of the future remnant liver, as compared both to PVE and LVD. Basing on previously published studies following success rates (as percentage of patients completing the second stage of treatment, the hepatic resection) have been assumed: 57% for PVE, 73% for LVD and 91% for ALPPS.

Assuming the thresholds for type I and type II error of 5% and 20% respectively, the calculated size of the study group should be 154 patients, more specifically 12 in the PVE group, 71 in the LVD group and 71 in the ALPPS group.

Special surveillance will be applied to patients in the PVE group and in case of low efficacy (<50%) in the first 6 patients, randomization to this group will be withheld.

Moreover, in case of unsuccessful induction of hypertrophy by the embolization techniques, patients may be qualified to rescue ALPPS procedure.

Primary end-point:

Percentage of patients with successful resection (patients, who gained sufficient increase of the FRL to proceed to the liver resection) with no post-surgical 90-day mortality.

Secondary end-points:

1. the rate and degree of volume increase in different groups
2. the rate and degree of functional increase in different groups
3. CCI index and complication rate >=3 degree according to the Clavien-Dindo classification after the first stage of treatment
4. CCI index and complication rate >=3 degree according to the Clavien-Dindo classification after the second stage of treatment
5. overall duration of hospital stay

Patient will be randomly assigned to the three study groups. All patients will undergo an abdominal contrast enhanced computed tomography and 99mTc-mebrofenin scintigraphy prior to the first stage of treatment. During the first stage of treatment, patients will undergo, according to their group:

1. Embolization of portal vein branch (PVE, portal vein embolization)
2. Embolization of both portal vein branch and hepatic vein (LVD, liver venous deprivation)
3. Partial ALPPS (Associating Liver Partition and Portal vein Ligation for Staged hepatectomy) - ligation of portal vein branch with partial liver transection, preferentially by laparoscopic technique

Computed tomography scans and scintigraphy will be repeated at day 7, 14 and 21 after the first stage of treatment. The second stage of treatment, the liver resection, will be performed after achievement of sufficient mebrofenin clearance rate (>=2,69%/min/m2). In case of failure to reach the desired clearance rate, the measurements will be continued every 7 days up to date 42. In case of uncertainty and discrepancy between the volumetric assessment in the computed tomography scan and the mebrofenin scintigraphy, it will be allowed to proceed to stage two (partial hepatectomy) after joint consultation of at least 3 hepatobiliary surgeons, 1 radiologist and 1 nuclear medicine specialist.

Routine blood tests such as morphology, serum bilirubin and creatinine concentration, transaminase activity, gamma-glutamyltranspeptidase or INR will be performed according to the standard procedure in the Department of Liver, Transplant and General Surgery, namely at day 0 and 1 and every 2-3 days or more frequent in the next days, depending on the patient clinical status. An additional blood sample will be collected from patients (after receiving and additional informed consent from the patient) and will be stored in the biobank (according to "Quality Standards for Polish Biobanks" v.2.00). The samples will be stored at the LBBK biobank at Medical University of Warsaw.

All patients will be monitored for surgical and 90-day complications. The volume increase after first stage of treatment, the functional increase after first stage of treatment, percentage of patients successfully proceeding to the second stage of treatment and complication rate will be calculated.

The percentage of patients with complications >= 3 degree in Clavien-Dindo classification and CCI index for each patient will be calculated.

Furthermore, the blood test results will be assessed to search for associations with patients' outcomes. Any possible differences in terms of baseline patients characteristics between groups will be addressed.

Statistical analysis will be performed using U Mann-Whitney test, exact Fisher's test, logistic regression, general linear models, Kaplan-Meier method and log-rank test. All three groups will be assessed in terms of occurrence of primary and secondary end-points.

The study is designed to last 6 years, from 1st June 2023 to 31st May 2029. The firsts four months are planned for the initiation of the study, the following months for recruitment, intervention and observation and the last two months for analyzing the results.

After discharge from the hospital, 2 control visit will be scheduled for each patient, 30 and 90 days after the liver resection. Further treatment will be continued in local oncological centers.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* patients qualified for liver resection
* future remnant liver <30% of standard liver volume
* written informed consent

Exclusion Criteria:

* liver cirrhosis
* pregnancy
* poor general health status or comorbidities excluding general anesthesia or hepatic resection
* contraindications to iodine contrast agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Successful resection | 6 months
  Percentage of patients with successful resection (patients, who gained sufficient increase of the FRL to proceed to the liver resection) with no post-surgical 90-day mortality.

SECONDARY OUTCOMES:
Change in future liver remnant volume over time | 42 days
  The rate of future liver remnant volume change (cm3/day) in different groups, assessed on computed tomography scans
Total relative change of future liver remnant volume | 42 days
  The degree (%) of volume increase in different groups, assessed on computed tomography scans
Change in future liver remnant functional capacity over time | 42 days
  The rate of functional increase (%/min/m2/day) in different groups, assessed on 99mTc-mebrofenin scintigraphy
Total relative change in future liver remnant functional capacity | 42 days
  The degree (%) of functional increase in different groups, assessed on 99mTc-mebrofenin scintigraphy
Severe morbidity after the first stage of treatment | 90 days
  Development of any complication >=3 degree according to the Clavien-Dindo classification after the first stage of treatment (censored at completion of the second stage or 90days)
Cumulative morbidity after the first stage of treatment | 90 days
  Comprehensive Complication Index after the first stage of treatment (censored at completion of the second stage or 90days)
Severe morbidity after the second stage of treatment | 90 days
  Development of any complication >=3 degree according to the Clavien-Dindo classification after the second stage of treatment
Cumulative morbidity after the second stage of treatment | 90 days
  Comprehensive Complication Index after the second stage of treatment
Overall morbidity | 1 year
  Overall duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Grąt, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Second Department of Clinical Radiology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be shared by the principal Investigator upon reasonable request.